CLINICAL TRIAL: NCT01598935
Title: Double Blind Controlled Trial of Protein in Active Children
Brief Title: Post-exercise Protein Intake for Active Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Nestec Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 10.44.NRC
Record Dates: First submitted 2012-02-16; First posted 2012-05-15 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Child
MeSH Terms: interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Placebo Comparator): placebo
  Interventions: Other: nutrition
- High protein intake (Active Comparator): Nutrition - High protein
  Interventions: Other: nutrition
- Low protein intake (Active Comparator): Nutrition - Low protein
  Interventions: Other: nutrition
- Medium protein intake (Active Comparator): Nutrition - Medium protein
  Interventions: Other: nutrition

INTERVENTIONS:
Other: nutrition — protein-based food

SUMMARY:
Today, there is an important lack of knowledge on the effects of dietary protein on protein metabolism after physical activity in children. Here, the investigators will measure changes in whole body protein metabolism using minimally invasive techniques and stable isotope methodology at rest and after physical activity with the intake of milk protein.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and physically active (as determined by medical and activity questionnaire)
* 10-12 years of age
* Within approximately 2 years of estimated age of peak height velocity (PHV)
* Minimum aerobic fitness of 35 ml/kg/min as assessed by the McMaster All-out Progressive Continuous Cycling Protocol
* Having obtained his/her informed assent
* Having obtained his/her legal representative's informed consent

Exclusion Criteria:

* Post-pubertal
* Taking any medication
* Smoker
* Undergoing medical treatment or investigations
* Body mass index > 24
* Suffer from chronic diseases (with regular intake of drugs, medical history)
* Vegetarians
* Vaccination in the last 4 months
* Any know food allergies or intolerance
* Pregnancy
* Special diet or weight loss program (e.g. Atkins diet)
* Acute illness
* Fever, cold, flu
* Participation in a cholesterol management program with functional foods like food supplement enriched in omega-3 fatty acids, dairy products enriched with phytosterols (margarines, yoghurts).

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2011-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Whole body protein balance | Participants will be followed for 10 days prior to assessment of whole body protein balance.
  Whole body protein balance will be measured by stable isotopes.

SECONDARY OUTCOMES:
Whole body protein metabolism, metabolites | Participants will be followed for 10 days prior to assessment of whole body protein metabolism and metabolites
  Whole body protein metabolism by stable isotopes and metabolite concentrations in plasma and urine.

CONTACTS AND LOCATIONS:
Overall Officials: Brian W Timmons, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Volterman KA, Moore DR, Breithaupt P, Godin JP, Karagounis LG, Offord EA, Timmons BW. Postexercise Dietary Protein Ingestion Increases Whole-Body Leucine Balance in a Dose-Dependent Manner in Healthy Children. J Nutr. 2017 May;147(5):807-815. doi: 10.3945/jn.116.239756. Epub 2017 Apr 5. PMID 28381530